CLINICAL TRIAL: NCT03113032
Title: Novel Pre-Surgery Exercise-Conditioning in Patients Waiting for Total Knee Arthroplasty (TKA)
Acronym: P-SEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Collaborators: Queen Margaret University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P-SEC001
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2017-06

CONDITIONS: Osteo Arthritis Knee
Keywords: total knee replacement; sensorimotor training; pre-surgery exercise; sensorimotor function; neuromuscular

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Feasibility Study
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The chief investigator who will deliver the exercise protocol will be blinded as to which leg is the intended leg for surgery. This will be done by another member of the medical team allocating the patients in block randomisation as they come in from the waiting list. This list with the respective "surgical" leg will be kept safely away from the chief investigator until all data is recorded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise group 1 (Experimental): This group of patients will receive the P-SEC exercise intervention protocol on their 'surgical' leg in addition to their normal pre-surgical care.
  Interventions: Other: P-SEC Pre-Surgical Care
- Exercise group 2 (Experimental): This group of patients will receive the P-SEC exercise intervention protocol on their 'non-surgical' leg in addition to their normal pre-surgical care.
  Interventions: Other: P-SEC Pre-Surgical Care
- Control group (Active Comparator): This group of patients will not receive the P-SEC protocol but will follow normal pre-surgical care along with the other two groups of patients.
  Interventions: Other: Normal pre-surgical care

INTERVENTIONS:
Other: P-SEC Pre-Surgical Care — The P-SEC protocol is designed to deliver a focal mode of exercise-conditioning for motor performance to the knee extensor musculature. The latter requires a brief, machine-based gravity-resisted joint' movements (<2 seconds). An exercise session (6-minutes, approximately) will require a patient to undertake 4 sets of movement, with sets separated by 60-seconds recovery (delivering a total of 36 exercises across 3 interspersed days).
  Arms: Exercise group 1; Exercise group 2
Other: Normal pre-surgical care — Routine pre-surgical care
  Arms: Control group

SUMMARY:
Total knee replacement (TKR) is the treatment of choice for patients suffering from long standing severe pain, functional limitation and instability caused by osteoarthritis (OA) of the knee joint's surfaces. Long standing arthritic joint surfaces, more often lead to pain and swelling and other physical factors that may contribute to knee joint instability. This instability causes a feeling of 'unsteadiness' whilst walking and may also contribute to falls. In view of the latter, it is important for this issue of 'unsteadiness' to be addressed. TKR helps to remove the cause of pain and swelling, but exercises are crucial to counteract the joint' instability and any feeling of 'unsteadiness' before and after surgery. However, research hasn't yet identified the optimum approach for delivering exercises that will help in patients' rehabilitation. Current studies have tried to incorporate rehabilitation programmes to improve this issue, but required a delivery of 6-8 weeks of exercises which has resulted in a logistical burden in view of the long duration. We have scientifically developed a new programme of exercise for the muscles of the knee that can be delivered during a single week prior to surgery. The pre-surgery exercise-programme (P-SEC), potentially offers similar effectiveness for improving the feeling of 'unsteadiness' and muscle' fitness as programmes that last much longer. Therefore, the purpose of this research study is to test the effectiveness of this new, short approach to exercising in patients who are waiting for a TKR surgery.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is the treatment of choice for patients suffering from severe pain and functional limitation caused by osteoarthritis (OA) of the knee joint's surfaces (Magee et al. 2009). Within the UK, over 60,000 TKA surgeries are registered yearly (NJR 2015), making TKA one of the most common surgeries of the joint. Rehabilitation following surgery is essential for recovery and with TKA this is crucial in regaining movement, function and control. Current rehabilitation mainly focuses on post-surgery rehabilitation to increase range of motion (ROM) and muscle power, and to aid in achieving a quick return to functional independence for patients. Despite this, research has shown that patients undergoing TKA, still continue to experience reduced capacities in neuromuscular responses which are required for quick knee joint reactions, stability and proprioception, up to months following TKA surgery (Silva et al. 2003). A deficit in an individual's knee joint proprioception (synonymously referred to as a deficit in sensorimotor performance), together with impaired strength, can lead to reduced functional balance capabilities and movement control (Piva et al. 2010; Rätsepsoo et al. 2011), and can also contribute to injury (Lephart et al. 1997) and a greater risk of falls (Swinkels et al. 2009; Bade et al. 2010; Rätsepsoo et al. 2011). In part, the latter may be due to time-constraints within the health-care system, where a necessary preservation of the primary focus, to decrease pain and improve general function in patients following a TKA, has sometimes been to the detriment of other aspects of rehabilitation.

Pre-surgery exercise-conditioning:

Studies have investigated the effects of pre-surgery exercise' (also known as pre-habilitation exercise) interventions on strength and sensorimotor performance deficits in patients undergoing TKA, through various modes of exercise. Their aim has been to utilise a period of time pre-surgery to improve patients' rehabilitation status (Huber et al. 2015; Topp et al. 2009; Desmueles et al. 2013; Mackay et al. 2012). However, the patterns of patients' adaptations to the generic exercise stimuli used within these studies, has not shown the gains that had been expected by physiological dose-response, and ultimately questioned the efficacy of using pre-habilitation for effective gains in long-term outcomes. Nevertheless, the concept of achieving early gains to conditioning status that might potentiate patients' later rehabilitation processes and status, remains attractive to the latter (Calatayud et al. 2016, Huber et al. 2015) and the NHS (Rooks et al. 2006; Crowe and Henderson, 2003).

Conditioning for enhanced sensorimotor performance has been consistently endorsed in the sports-medical and sports-performance (Hubscher et al. 2010; Mandelbaum et al. 2005) and clinical literature (Tsao et al. 2007; Granacher et al. 2006) for its causal relationship to reduced injury likelihood and capability to improve function. While the precise dose of stimuli to achieve gains in sensorimotor performance is less clearly defined, enhancing motor performance by means of exercise that resist the effects of gravity or externally-applied loading to a joint system, has established underpinnings physiologically by improving motor performance and indirectly effecting sensorimotor responses (Vikne et al. 2006; Hakan et al. 2002; Moran et al. 2007). Clinically, the challenge has been to formulate a suitably pragmatic programme of conditioning that will accommodate the time- and cost-pressures associated with contemporary care practice while simultaneously offering efficacy when delivered prior to surgery as a pre-habilitative intervention. Rehabilitative and prophylactic conditioning programmes used in current studies for enhanced neuromuscular and sensorimotor performance, have typically required and been delivered in a duration of 6-8-weeks (Calatayud et al. 2016; Huber et al. 2015; Topp et al. 2009; Desmueles et al. 2013; Mackay et al. 2012). This has commanded a substantive logistical burden to elicit expected gains.

A novel approach to conditioning - Development of the P-SEC protocol:

A novel formulation of conditioning that could condense the pattern of delivery of physiologically-effective, dose-related stimuli, while simultaneously maintaining the vast proportion of potential gains in performance, would offer advantages to patients and clinicians for logistical versatility with which a package of conditioning might be delivered. This would be especially important within the relatively short period of time between the patients electing for surgery after clinical consultation and a surgical procedure, if pre-habilitation were to be incorporated effectively within care pathways. Recent studies have shown that with careful periodization and micro-cyclical management of the mode of exercise-conditioning, patterning of exercise intensity and work/recovery ratios, and progression of increasing physiological stimuli for adaptation, it is possible to deliver gains in neuromuscular performance within a programme lasting 2-3-weeks, which match 70% of the effects expected during longer programmes (Peer and Gleeson, in press; Peer et al. under review). Additional adaptations to this intervention model would be needed to counteract arthrogenic and autogenic sources of inhibition associated with long-term disease conditions such as OA (Rice et al. 2010), limiting neuromuscular performance and conditioning gains by the intrusion of nociceptive stimuli such as an increase in intra-articular joint pressure (Palmieri-Smith et al. 2007). The cost-neutrality of the embedding pre-habilitative conditioning for improved motor performance might be feasible if a portion of the end-phase rehabilitation following a surgical procedure, which has been shown recently to offer limited gains in performance within the formal care pathway (Bailey et al. 2014), could be sacrificed in favour of an equivalent time- period of conditioning prior to surgery.

Therefore, the purpose of the P-SEC study is to undertake a randomized controlled feasibility trial in order to investigate the effects of this new formulation of exercise-conditioning for motor performance on objectively-measured and patient-perceived sensorimotor, functional and psychophysiological performance capacities in patients waiting for a TKA.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females over the age of 18, diagnosed with severe osteoarthritis (OA) of the knee and awaiting a TKA (Including contralateral knee OA/TKA and/or other orthopaedic conditions affecting the contralateral leg)

Exclusion Criteria:

* Individuals undertaking TKA due to a knee joint disease other than osteoarthritis
* Rheumatic disorder
* Neurological disorders
* Other orthopaedic conditions affecting lower body function
* Individuals with reduced mental capacity affecting their ability to follow exercise programme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Electromechanical delay (EMD) | 11 months
  The primary outcome measure for this study is the measurement of Electromechanical Delay (EMD) of the knee extensor musculature. The data obtained will give an indication of the participants' sensorimotor and neuromuscular performance capacities. Measurements of the latter's activity will be obtained from electromechanical signals collected by a purpose built dynamometer (Gleeson et al. 2013) and EMG signals obtained from surface electrodes over the knee extensor musculature.

SECONDARY OUTCOMES:
Balance Force plate | 11 months
  Measurement of postural control indices through the use of a standing balance force plate
Peak Force (PF) | 11 months
  Further measurements of Sensorimotor and Neuromuscular performance capacities using data obtained from the EMG and seated dynamometer used for the primary outcome measurement.
Rate of force Development (RFD) | 11 months
  Further measurements of Sensorimotor and Neuromuscular performance capacities using data obtained from the EMG and seated dynamometer used for the primary outcome measurement.
Knee Injury and Osteoarthritis questionnaire (KOOS) questionnaire | 11 months
  Subjective measurement of patients' performance capacity
Oxford Knee score (OKS) | 11 months
  Subjective measurement of patients' performance capacity
Performance profile questionnaire | 11 months
  Subjective measurement of patients' performance capacity
Pain self efficacy questionnaire | 11 months
  Subjective measurement of patients' performance capacity
Short Form Health Questionnaire (SF36v2) | 11 months
  Subjective measurement of patients' performance capacity
International Physical Activity Questionnaire (IPAQ) | 11 months
  Subjective measurement of patients' performance capacity

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Gleeson, Prof., Study Director — Queen Margaret University; Anna Maria Risso, Ms, Principal Investigator — Queen Margaret University
Locations (1):
- Robert Jones and Agnes Hunt NHS Trust Foundation, Oswestry, Gobowen, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Risso AM, van der Linden ML, Bailey A, Gallacher P, Gleeson N. Exploratory insights into novel prehabilitative neuromuscular exercise-conditioning in total knee arthroplasty. BMC Musculoskelet Disord. 2022 Jun 7;23(1):547. doi: 10.1186/s12891-022-05444-0. PMID 35672761